CLINICAL TRIAL: NCT06182956
Title: Evaluation of Physiological Effects of Noninvasive Mechanical Ventilation and High-flow Oxygen Therapy for Acute Exacerbations of Interstitial Lung Diseases
Brief Title: NIV Versus HFO for Acute Exacerbations of Interstitial Lung Diseases
Acronym: IRAPIDPhysio
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRAPIDPhysio
Record Dates: First submitted 2023-08-22; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Interstitial Lung Disease; Acute Respiratory Failure
Keywords: Noninvasive mechanical ventilation; Nasal high-flow oxygen therapy; Respiratory work; Hemodynamics; Diaphragm
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- NIV + CPAP + HFO (Experimental): The patient will be placed under noninvasive mechanical ventilation during 30 min, then continuous positive airway pressure during 30 min and then nasal high-flow oxygen during 30 min. Each period will be separated by a washout period of maximum 30 min under oxygen with a non-rebreathing mask.
  Interventions: Device: Noninvasive mechanical ventilation; Device: Nasal high-flow oxygen therapy; Device: Continuous positive airway pressure
- NIV + HFO + CPAP (Experimental): The patient will be placed under noninvasive mechanical ventilation during 30 min, then nasal high-flow oxygen during 30 min and then continuous positive airway pressure during 30 min. Each period will be separated by a washout period of maximum 30 min under oxygen with a non-rebreathing mask.
  Interventions: Device: Noninvasive mechanical ventilation; Device: Nasal high-flow oxygen therapy; Device: Continuous positive airway pressure
- CPAP + NIV + HFO (Experimental): The patient will be placed under continuous positive airway pressure during 30 min, then noninvasive mechanical ventilation during 30 min and then nasal high-flow oxygen during 30 min. Each period will be separated by a washout period of maximum 30 min under oxygen with a non-rebreathing mask.
  Interventions: Device: Noninvasive mechanical ventilation; Device: Nasal high-flow oxygen therapy; Device: Continuous positive airway pressure
- CPAP + HFO + NIV (Experimental): The patient will be placed under continuous positive airway pressure during 30 min, then nasal high-flow oxygen during 30 min and then noninvasive mechanical ventilation during 30 min. Each period will be separated by a washout period of maximum 30 min under oxygen with a non-rebreathing mask.
  Interventions: Device: Noninvasive mechanical ventilation; Device: Nasal high-flow oxygen therapy; Device: Continuous positive airway pressure
- HFO + CPAP + NIV (Experimental): The patient will be placed under nasal high-flow oxygen during 30 min, then continuous positive airway pressure during 30 min and then noninvasive mechanical ventilation during 30 min. Each period will be separated by a washout period of maximum 30 min under oxygen with a non-rebreathing mask.
  Interventions: Device: Noninvasive mechanical ventilation; Device: Nasal high-flow oxygen therapy; Device: Continuous positive airway pressure
- HFO + NIV + CPAP (Experimental): The patient will be placed under nasal high-flow oxygen during 30 min, then noninvasive mechanical ventilation during 30 min and then continuous positive airway pressure during 30 min. Each period will be separated by a washout period of maximum 30 min under oxygen with a non-rebreathing mask.
  Interventions: Device: Noninvasive mechanical ventilation; Device: Nasal high-flow oxygen therapy; Device: Continuous positive airway pressure

INTERVENTIONS:
Device: Noninvasive mechanical ventilation — Noninvasive mechanical ventilation is a respiratory technique which allows the administration of positive inspiratory and expiratory airway pressures in order to ventilate the lungs.
Device: Nasal high-flow oxygen therapy — Nasal high-flow is a respiratory technique which allows the administration of warmed and humidified air, associated with oxygen.
Device: Continuous positive airway pressure — Continuous positive airway pressure is a respiratory technique which allows to maintain a constant positive airway pressure during inspiration and expiration.

SUMMARY:
The objectives of this study are to compare the physiological consequences of high-flow oxygen therapy and noninvasive mechanical ventilation on ventilation, respiratory work and hemodynamics during acute respiratory failure in diffuse interstitial pneumonia.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 yrs
* Hospitalization in intensive care unit
* Acute exacerbation of a previously/presently documented diffuse (fibrotic) interstitial lung disease
* Dyspnea majoration since at least 1 month
* Alveolar or ground-glass opacities on CT-scan that are superposed to interstitial lung disease and not explained by left heart failure or volume overload
* Hypoxemia requiring oxygen flows > 6 L/min

Exclusion criteria:

* Contraindication to noninvasive ventilation or high-flow oxygen therapy
* Immediate indication to endotracheal intubation or hemodynamic assistance
* Body mass index > 40
* Presence of a pacemaker or an implantable defibrillator
* Presence of cutaneous lesions where Pulmovista® belt should be placed
* Moribund patient
* Pregnant or breastfeeding women or women of childbearing age without an effective method of contraception
* Protected adult patient (tutorship or curatorship)
* Patient deprived of liberty by court or administrative decision
* No possibility to install nasogastric tube
* Endotracheal or tracheostomy tube requirement during the study
* Hemodynamic assistance requirement during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary compliance | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of global pulmonary compliance (Cglob) under noninvasive ventilation (NIV) and high-flow oxygen therapy (HFO) during acute respiratory failure in diffuse interstitial pneumonia.

SECONDARY OUTCOMES:
Pulmonary compliance | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of global pulmonary compliance (Cglob) under NIV and continuous positive airway pressure (CPAP) during acute respiratory failure in diffuse interstitial pneumonia.
Pulmonary compliance | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of global pulmonary compliance (Cglob) under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
Pulmonary compliance | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of global pulmonary compliance (Cglob) under HFO and face mask oxygen therapy (FM) during acute respiratory failure in diffuse interstitial pneumonia.
Pulmonary compliance | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of global pulmonary compliance (Cglob) under NIV and face mask oxygen therapy (FM) during acute respiratory failure in diffuse interstitial pneumonia.
Pulmonary compliance | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of global pulmonary compliance (Cglob) under CPAP and face mask oxygen therapy (FM) during acute respiratory failure in diffuse interstitial pneumonia.
Tidal volume | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Tidal volume under CPAP and face mask oxygen therapy (FM) during acute respiratory failure in diffuse interstitial pneumonia.
Tidal volume | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Tidal volume under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
Tidal volume | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Tidal volume under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
Tidal volume | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Tidal volume under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.
Tidal volume | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Tidal volume under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
Tidal volume | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Tidal volume under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
end-expiratory lung volume | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of end-expiratory lung volume under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
end-expiratory lung volume | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of end-expiratory lung volume under NIV and HFO during acute respiratory failure in diffuse interstitial pneumonia.
end-expiratory lung volume | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of end-expiratory lung volume under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
end-expiratory lung volume | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of end-expiratory lung volume under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
end-expiratory lung volume | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of end-expiratory lung volume under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
end-expiratory lung volume | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of end-expiratory lung volume under FM and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
transpulmonary pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transpulmonary pressure under FM and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
transpulmonary pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transpulmonary pressure under FM and HFO during acute respiratory failure in diffuse interstitial pneumonia.
transpulmonary pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transpulmonary pressure under FM and NIV during acute respiratory failure in diffuse interstitial pneumonia.
transpulmonary pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transpulmonary pressure under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.
transpulmonary pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transpulmonary pressure under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
transpulmonary pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transpulmonary pressure under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
driving pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of driving pressure under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
driving pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of driving pressure under NIV and HFO during acute respiratory failure in diffuse interstitial pneumonia.
driving pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of driving pressure under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
driving pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of driving pressure under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
driving pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of driving pressure under CPAP and HFO during acute respiratory failure in diffuse interstitial pneumonia.
driving pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of driving pressure under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
Global inhomogeneity index | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Global inhomogeneity index under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
Global inhomogeneity index | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Global inhomogeneity index under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
Global inhomogeneity index | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Global inhomogeneity index under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
Global inhomogeneity index | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Global inhomogeneity index under NIV and HFO during acute respiratory failure in diffuse interstitial pneumonia.
Global inhomogeneity index | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Global inhomogeneity index under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
Global inhomogeneity index | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Global inhomogeneity index under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
respiratory rate | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of respiratory rate under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
respiratory rate | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of respiratory rate under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.
respiratory rate | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of respiratory rate under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
respiratory rate | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of respiratory rate under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
respiratory rate | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of respiratory rate under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
respiratory rate | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of respiratory rate under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
inspiratory time | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of inspiratory time under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
inspiratory time | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of inspiratory time under NIV and HFO during acute respiratory failure in diffuse interstitial pneumonia.
inspiratory time | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of inspiratory time under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
inspiratory time | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of inspiratory time under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
inspiratory time | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of inspiratory time under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
inspiratory time | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of inspiratory time under CPAP and NIV during acute respiratory failure in diffuse interstitial pneumonia.
inspiratory time | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of inspiratory time under CPAP and HFO during acute respiratory failure in diffuse interstitial pneumonia.
oesophagal pressure swings | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of oesophagal pressure variations between inspiration and expiration under CPAP and HFO during acute respiratory failure in diffuse interstitial pneumonia.
oesophagal pressure swings | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of oesophagal pressure variations between inspiration and expiration under CPAP and NIV during acute respiratory failure in diffuse interstitial pneumonia.
oesophagal pressure swings | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of oesophagal pressure variations between inspiration and expiration under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
oesophagal pressure swings | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of oesophagal pressure variations between inspiration and expiration under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
oesophagal pressure swings | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of oesophagal pressure variations between inspiration and expiration under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
oesophagal pressure swings | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of oesophagal pressure variations between inspiration and expiration under NIV and HFO during acute respiratory failure in diffuse interstitial pneumonia.
transdiaphragmatic pressure variations | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transdiaphragmatic pressure variations between inspiration and expiration under NIV and HFO during acute respiratory failure in diffuse interstitial pneumonia.
transdiaphragmatic pressure variations | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transdiaphragmatic pressure variations between inspiration and expiration under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
transdiaphragmatic pressure variations | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transdiaphragmatic pressure variations between inspiration and expiration under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
transdiaphragmatic pressure variations | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transdiaphragmatic pressure variations between inspiration and expiration under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
transdiaphragmatic pressure variations | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transdiaphragmatic pressure variations between inspiration and expiration under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
transdiaphragmatic pressure variations | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transdiaphragmatic pressure variations between inspiration and expiration under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
transdiaphragmatic pressure time products | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transdiaphragmatic pressure time products under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
transdiaphragmatic pressure time products | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transdiaphragmatic pressure time products under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.
transdiaphragmatic pressure time products | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transdiaphragmatic pressure time products under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
transdiaphragmatic pressure time products | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transdiaphragmatic pressure time products under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
transdiaphragmatic pressure time products | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transdiaphragmatic pressure time products under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
transdiaphragmatic pressure time products | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transdiaphragmatic pressure time products under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
oesophagal pressure time products | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of oesophagal pressure time products under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
oesophagal pressure time products | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of oesophagal pressure time products under NIV and HFO during acute respiratory failure in diffuse interstitial pneumonia.
oesophagal pressure time products | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of oesophagal pressure time products under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
oesophagal pressure time products | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of oesophagal pressure time products under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
oesophagal pressure time products | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of oesophagal pressure time products under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
oesophagal pressure time products | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of oesophagal pressure time products under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
ultrasound diaphragmatic strain. | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of ultrasound diaphragmatic strain under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
diaphragmatic thickening fraction | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of diaphragmatic thickening fraction under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
diaphragmatic thickening fraction | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of diaphragmatic thickening fraction under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.
diaphragmatic thickening fraction | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of diaphragmatic thickening fraction under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
diaphragmatic thickening fraction | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of diaphragmatic thickening fraction under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
diaphragmatic thickening fraction | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of diaphragmatic thickening fraction under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
diaphragmatic thickening fraction | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of diaphragmatic thickening fraction under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
peak inspiratory flow | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of peak inspiratory flow under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
peak inspiratory flow | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of peak inspiratory flow under NIV and HFO during acute respiratory failure in diffuse interstitial pneumonia.
peak inspiratory flow | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of peak inspiratory flow under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
peak inspiratory flow | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of peak inspiratory flow under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
peak inspiratory flow | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of peak inspiratory flow under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
peak inspiratory flow | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of peak inspiratory flow under FM and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
peak expiratory flow | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of peak expiratory flow under FM and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
peak expiratory flow | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of peak expiratory flow under FM and NIV during acute respiratory failure in diffuse interstitial pneumonia.
peak expiratory flow | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of peak expiratory flow under FM and HFO during acute respiratory failure in diffuse interstitial pneumonia.
peak expiratory flow | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of peak expiratory flow under CPAP and HFO during acute respiratory failure in diffuse interstitial pneumonia.
peak expiratory flow | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of peak expiratory flow under CPAP and NIV during acute respiratory failure in diffuse interstitial pneumonia.
peak expiratory flow | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of peak expiratory flow under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.
Systolic arterial pressures | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Systolic arterial pressures under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
Systolic arterial pressures | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Systolic arterial pressures under NIV and HFO during acute respiratory failure in diffuse interstitial pneumonia.
Systolic arterial pressures | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Systolic arterial pressures under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
Systolic arterial pressures | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Systolic arterial pressures under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
Systolic arterial pressures | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Systolic arterial pressures under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
Systolic arterial pressures | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Systolic arterial pressures under CPAP and HFO during acute respiratory failure in diffuse interstitial pneumonia.
Diastolic arterial pressures | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Diastolic arterial pressures under CPAP and HFO during acute respiratory failure in diffuse interstitial pneumonia.
Diastolic arterial pressures | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Diastolic arterial pressures under CPAP and NIV during acute respiratory failure in diffuse interstitial pneumonia.
Diastolic arterial pressures | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Diastolic arterial pressures under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
Diastolic arterial pressures | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Diastolic arterial pressures under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
Diastolic arterial pressures | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Diastolic arterial pressures under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
Diastolic arterial pressures | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Diastolic arterial pressures under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.
Mean arterial pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Mean arterial pressures under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.
Mean arterial pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Mean arterial pressures under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
Mean arterial pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Mean arterial pressures under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
Mean arterial pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Mean arterial pressures under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
Mean arterial pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Mean arterial pressures under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
Mean arterial pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Mean arterial pressures under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
systolic pulmonary arterial pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of systolic pulmonary arterial pressure under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
systolic pulmonary arterial pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of systolic pulmonary arterial pressure under NIV and HFO during acute respiratory failure in diffuse interstitial pneumonia.
systolic pulmonary arterial pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of systolic pulmonary arterial pressure under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
systolic pulmonary arterial pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of systolic pulmonary arterial pressure under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
systolic pulmonary arterial pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of systolic pulmonary arterial pressure under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
systolic pulmonary arterial pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of systolic pulmonary arterial pressure under CPAP and NIV during acute respiratory failure in diffuse interstitial pneumonia.
tricuspid annular plane systolic excursion | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of tricuspid annular plane systolic excursion under CPAP and NIV during acute respiratory failure in diffuse interstitial pneumonia.
tricuspid annular plane systolic excursion | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of tricuspid annular plane systolic excursion under CPAP and HFO during acute respiratory failure in diffuse interstitial pneumonia.
tricuspid annular plane systolic excursion | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of tricuspid annular plane systolic excursion under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
tricuspid annular plane systolic excursion | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of tricuspid annular plane systolic excursion under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
tricuspid annular plane systolic excursion | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of tricuspid annular plane systolic excursion under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
tricuspid annular plane systolic excursion | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of tricuspid annular plane systolic excursion under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.
right ventricular strain | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of right ventricular strain under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.
right ventricular strain | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of right ventricular strain under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
right ventricular strain | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of right ventricular strain under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
right ventricular strain | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of right ventricular strain under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
right ventricular strain | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of right ventricular strain under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
right ventricular strain | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of right ventricular strain under CPAP and NIV during acute respiratory failure in diffuse interstitial pneumonia.
left ventricular ejection fraction | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of left ventricular ejection fraction under CPAP and NIV during acute respiratory failure in diffuse interstitial pneumonia.
left ventricular ejection fraction | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of left ventricular ejection fraction under CPAP and HFO during acute respiratory failure in diffuse interstitial pneumonia.
left ventricular ejection fraction | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of left ventricular ejection fraction under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
left ventricular ejection fraction | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of left ventricular ejection fraction under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
left ventricular ejection fraction | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of left ventricular ejection fraction under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
left ventricular ejection fraction | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of left ventricular ejection fraction under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.
E/E' ratio | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of E/E' ratio under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.
E/E' ratio | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of E/E' ratio under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
E/E' ratio | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of E/E' ratio under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
E/E' ratio | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of E/E' ratio under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
E/E' ratio | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of E/E' ratio under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
E/E' ratio | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of E/E' ratio under CPAP and NIV during acute respiratory failure in diffuse interstitial pneumonia.
right auricular pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of right auricular pressure under CPAP and NIV during acute respiratory failure in diffuse interstitial pneumonia.
right auricular pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of right auricular pressure under CPAP and HFO during acute respiratory failure in diffuse interstitial pneumonia.
right auricular pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of right auricular pressure under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
right auricular pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of right auricular pressure under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
right auricular pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of right auricular pressure under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
right auricular pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of right auricular pressure under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.
cardiac output | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of cardiac output under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.
cardiac output | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of cardiac output under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
cardiac output | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of cardiac output under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
cardiac output | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of cardiac output under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
cardiac output | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of cardiac output under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
cardiac output | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of cardiac output under CPAP and NIV during acute respiratory failure in diffuse interstitial pneumonia.
heart rate | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of heart rate under CPAP and NIV during acute respiratory failure in diffuse interstitial pneumonia.
heart rate | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of heart rate under CPAP and HFO during acute respiratory failure in diffuse interstitial pneumonia.
heart rate | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of heart rate under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
heart rate | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of heart rate under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
heart rate | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of heart rate under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
heart rate | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of heart rate under NIV and HFO during acute respiratory failure in diffuse interstitial pneumonia.
Pulsed oxymetry | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of pulsed oxymetry under NIV and HFO during acute respiratory failure in diffuse interstitial pneumonia.
Pulsed oxymetry | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of pulsed oxymetry under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
Pulsed oxymetry | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of pulsed oxymetry under NIV and FM during acute respiratory failure in diffuse interstitial pneumonia.
Pulsed oxymetry | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of pulsed oxymetry under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
Pulsed oxymetry | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of pulsed oxymetry under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
Pulsed oxymetry | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of pulsed oxymetry under CPAP and HFO during acute respiratory failure in diffuse interstitial pneumonia.
transcutaneous carbon dioxide pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transcutaneous carbon dioxide pressure under CPAP and HFO during acute respiratory failure in diffuse interstitial pneumonia.
transcutaneous carbon dioxide pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transcutaneous carbon dioxide pressure under CPAP and FM during acute respiratory failure in diffuse interstitial pneumonia.
transcutaneous carbon dioxide pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transcutaneous carbon dioxide pressure under CPAP and NIV during acute respiratory failure in diffuse interstitial pneumonia.
transcutaneous carbon dioxide pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transcutaneous carbon dioxide pressure under FM and NIV during acute respiratory failure in diffuse interstitial pneumonia.
transcutaneous carbon dioxide pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transcutaneous carbon dioxide pressure under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.
transcutaneous carbon dioxide pressure | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of transcutaneous carbon dioxide pressure under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
Dyspnea | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Borg's scale (from 0 to 10, 10 is maximal dyspnea) under HFO and FM during acute respiratory failure in diffuse interstitial pneumonia.
Dyspnea | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Borg's scale (from 0 to 10, 10 is maximal dyspnea) under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.
Dyspnea | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Borg's scale (from 0 to 10, 10 is maximal dyspnea) under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
Dyspnea | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Borg's scale (from 0 to 10, 10 is maximal dyspnea) under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
Dyspnea | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Borg's scale (from 0 to 10, 10 is maximal dyspnea) under FM and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
Dyspnea | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Comparison of Borg's scale (from 0 to 10, 10 is maximal dyspnea) under FM and NIV during acute respiratory failure in diffuse interstitial pneumonia.
Comparison of Comfort | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Visual comfort scale (from 0 to 10, 10 is maximal confort) under FM and NIV during acute respiratory failure in diffuse interstitial pneumonia.
Comparison of Comfort | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Visual comfort scale (from 0 to 10, 10 is maximal confort) under FM and HFO during acute respiratory failure in diffuse interstitial pneumonia.
Comparison of Comfort | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Visual comfort scale (from 0 to 10, 10 is maximal confort) under FM and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
Comparison of Comfort | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Visual comfort scale (from 0 to 10, 10 is maximal confort) under NIV and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
Comparison of Comfort | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Visual comfort scale (from 0 to 10, 10 is maximal confort) under HFO and CPAP during acute respiratory failure in diffuse interstitial pneumonia.
Comparison of Comfort | During the intervention, after an exposure of 30 minutes to the oxygen therapy device
  Visual comfort scale (from 0 to 10, 10 is maximal confort) under HFO and NIV during acute respiratory failure in diffuse interstitial pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Elise ARTAUD-MACARI, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- ADIR Association, Rouen, France